CLINICAL TRIAL: NCT05987605
Title: A Phase I/II, First in Human, Single Arm, Open Label Study to Evaluate the Safety and Efficacy of the Injection of Triple-specific T-cell Engager 1A46in Adult Subjects with R/R CD20 Positive And/or CD19 Positive B Cell Non-Hodgkin's Lymphoma (B - NHL)
Brief Title: Phase I/II Clinical Study of 1A46 Drug Substance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor's Research and Development strategy adjustment
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BR110-I/II
Record Dates: First submitted 2023-07-10; First posted 2023-08-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1A46 Drug Substance (Experimental): One cycle is defined as 21 days. Patients will be scheduled to receive weekly infusions of 1A46 for the first cycle and then for the remaining 15 cycles of the study, patients will receive a single infusion of 1A46 per cycle (Q3W)
  Interventions: Drug: 1A46 Drug Substance

INTERVENTIONS:
Drug: 1A46 Drug Substance — Cycle 1 which will consist of an initial dose given on C1D1 and an intermediate dose given on C1D8, followed by a maintenance dose beginning on C1D15 and continuing while the patient is treated at that dose level

SUMMARY:
A phase I/II, first in human, single arm, open label study to evaluate the safety and efficacy of the injection of triple-specific T-cell engager 1A46 in adult subjects with R/R CD20 positive and/or CD19 positive B cell non-Hodgkin's lymphoma (B - NHL)

DETAILED DESCRIPTION:
This study is an open-label, multicenter, Phase 1 dose escalation and Phase 2 dose expansion study of 1A46 in adult patients with advanced relapsed/refractory (r/r) CD20 and/or CD19positive B-cell NHL for whom there is not available effective standard treatment . This study is the FIH study of 1A46 in China. This FIH study will include a dose escalation (Phase 1 part) and a dose expansion in 3 cohorts (Phase 2 part). If specific criteria for efficacy are met in one or more of the Phase 2 cohorts, a statistically validated number of additional patients will be enrolled with the goal of accelerated approval The starting dose for phase I is C1D1 1μg，C1D8 1μg，C1D15 and C2D1 afterwards 1 μg, followed by 10 dose cohorts. Duration of dose limiting toxicity (DLT) observation is 28 days.One cycle is defined as 21 days. Patients will be scheduled to receive weekly injection of 1A46 for the first cycles (3 weeks) and then for the remaining 15 cycles, the study patients will receive a single injection of 1A46 per cycle (every 3 weeks [Q3W]).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged 18 years or older; 2. Be able to sign informed consent form voluntarily and understand the study, incuding the purpose and the procedure and be able to comply with protocol requirements; 3. Patient populations:

Dose Escalation:

1. Aggressive NHL (aNHL) : MCL, each subtype of DLBCL and FL3b, PMBCL, high level of B cell lymphoma, etc.
2. Indolent NHL (iNHL) : including FL1-3 a grade, MZL, small lymphocytic lymphoma, etc.
3. all NHL patients should must: relapsed after or failed to respond to at least two prior systemic treatment regimens, including at least one containing an anti-CD20-directed therapy,, received or be ineligible for autologous SCT , there is no other standard treatment is thought to have clinical benefit

   Dose Expansion:

   Cohort 1: FL patients who are refractory to or relapsed after ≥ 2 prior regimens and have no other standard of care with clinical benefit.

   Cohort 2: r/r DLBCL patients who have progressed after or refractory to 2 or more lines of systemic therapy and have not received prior therapy with CAR-T, and do not have standard treatment with clinical benefit.

   Cohort 3: r/r DLBCL patients who have progressed after or refractory to 2 or more regimens which consisted of a CAR-T therapy that has been approved by a health authority, and do not have standard treatment with clinical benefit.

   4. NHL patients must have expression of CD20 and/or CD19-expression as determined by immunohistochemistry (IHC) at a certified laboratory within 6 months before study entry without intervening treatment of NHL, otherwise a fresh biopsy must be obtained to determine if CD19 and/or CD20 continue to be expressed by tumor cells.

   5. ≥ 1 measurable target lesion as defined by Lugano 2014 criteria (> 15 mm in its largest dimension for nodal lesions, or > 10 mm in its largest dimension for extranodal lesion).

   6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; Life expectancy> 3 months.

   7. Subjects with fertility must take effective contraceptive measures after signing the ICF until at least 12 months after the last administration of 1A46.

   8. Clinical laboratory values as specified below during the screening period.

   ① Total bilirubin must be < 1.5 x the upper limit of the normal range (ULN). Total bilirubin may be elevated up to 3 x ULN if their elevation can be reasonably ascribed to patients with documented Gilbert's Syndrome.
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be < 3 x ULN. AST and ALT may be elevated up to 5 x ULN if their elevation can be reasonably ascribed to the presence of metastatic disease in liver.

     * Calculated creatinine clearance > 50 mL/min (the Cockcroft-Gault formula). ④ Hemoglobin (Hb) must be ≥ 80 g/L. No transfusion of red blood cells or use of hematopoietic stimulating factors such as TPO within 14 days before the study.

       * Neutrophil count must be >1.0×10^9/L, No granulocyte or granulocyte macrophage colony-stimulating factor and other hematopoietic stimulating factors were used within 14 days before the study.

         * Platelet count must be >75×10^9/L, No platelet transfusion or use of hematopoietic stimulating factors such as TPO and IL-11 within 14 days prior to testing.

           ⑦ Prothrombin time-international normalized ratio (PT-INR) must be ≤ 1.5. Patients who are appropriately anticoagulated for a preexisting medical condition [e.g., atrial fibrillation] may be eligible with documented and evaluated by investigators and sponsor approval.

           9. Recovery to Grade 0-1 from AEs related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy.

   Exclusion Criteria:
   * 1. Patient has brain metastasis or other significant neurological conditions. 2. Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period, or intending to become pregnant during the study.

     3. At the time of enrollment, there are active infections, including bacteria, viruses (including EB virus, cytomegalovirus, etc.), fungi, mycobacteria, parasites, or other infections (excluding nail bed fungal infections), or there are any serious infections that require antibiotic intravenous injection treatment or hospitalization treatment (relating to the completion of the course of antibiotics) within the first 4 weeks prior to enrollment.

     4. Treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or immunosuppressive medication( including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs) ≤ 7 days before the first dose of 1A46, with the following exceptions: local, ocular, intra-articular, nasal, or inhaled corticosteroids, and those who receive corticosteroid replacement therapy due to adrenal insufficiency.

     5. Treatment with any investigational products (including cell or gene therapy) within 5 half-lives of the agent or 4 weeks prior to the first dose of 1A46, whichever is shorter.

     6. Received Systemic anticancer therapy (including I/O therapies) within 5 half-lives of the agent or 4 weeks prior to the first dose of 1A46, whichever is shorter.

     7. Treatment with radiotherapy within 2 weeks before the study entry. If the patients have received radiotherapy within 4 weeks before enrollment, there must be at least one measurable lesion outside the radiotherapy area, or if the patient only has measurable lesion progression after radiotherapy, they can be enrolled.

     8. Treatment with CAR-T within 30 days before the study entry. 9. Treatment with autologous stem cell transplantation therapy within 100 days before the study entry.

     10. Prior allogeneic hematopoietic stem cell transplantation . 11. Priorsolid organ transplantation. 12. Positive human immunodeficiency virus (HIV) antibodies; positive EB virus nucleic acid ; positive Cytomegalovirus nucleic acid positive; Hepatitis C virus (HCV) antibody is positive, and the result of HCV RNA detection is positive; Hepatitis B surface antigen [HBsAg] is positive, and hepatitis B virus DNA test result is positive or greater than the upper limit of normal value.

     13. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse. 14. Have ischemic or hemorrhagic cerebrovascular disease, epilepsy, dementia, or ≥ grade 3 gastrointestinal bleeding within the first 6 months (CTCAE, version 5.0) before screening.

     15. Unstable cardiovascular function:
     * Myocardial infarction occurred within 6 months prior to enrollment;

       * Have experienced unstable angina pectoris within 3 months prior to enrollment; ③ Uncontrolled and clinically significant arrhythmias (such as persistent ventricular tachycardia, ventricular fibrillation, and torsion of the apex);

         * Mobitz type II degree or III degree atrioventricular block; ⑤ Congestive heart failure with a New York Heart Association rating of ≥ 3; ⑥ Left ventricular ejection fraction<50%. 16. Received major surgery < 4 weeks prior to enrollment; (minor surgeries such as catheter insertion and biopsy required by the protocol are not considered as exclusion criteria).

           17. Inoculate with live virus vaccine within 28 days before enrollment (attenuated live vaccine is not allowed during the study period or until B cells return to normal range after the last trial drug administration).

           18. Have a history of grade 3-4 allergic reactions to other monoclonal antibody treatments; Or known to be allergic to any component or excipient of the investigational drug. Patients with Level 3 reactions lasting less than 24 hours may be eligible for inclusion after comprehensive evaluation by the researchers.

           19. Have a history of 3-4 levels of immune related adverse events or a history of immune related adverse events requiring discontinuation of medication, except for level 3 endocrine diseases treated with hormone replacement therapy. Subjects who have experienced levels 3-4 ICANS after previous CAR-T treatment.

           20. Any other serious underlying diseases that researchers believe may interfere with treatment, affect patient compliance, or put patients at high risk of treatment-related complications (such as active gastric ulcers, uncontrolled seizures, cerebrovascular events, gastrointestinal bleeding, severe signs and symptoms of coagulation disorders, heart disease), mental, psychological, familial, or geographic conditions.

           21. Have had other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell skin cancer.

           22. Autoimmune, liver, and lung diseases that may worsen under immune activation, such as certain autoimmune diseases, cirrhosis, hepatitis, interstitial pneumonia, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, multiple sclerosis, antiphospholipid antibody syndrome, vasculitis, psoriasis history, etc.

           23. Thoracic effusion, pericardial effusion, or ascites that require frequent drainage or medical intervention (recurrence within 2 weeks after intervention requires additional intervention).

           24. Previous T-cell engaging treatment regimens (including bispecific antibody, CAR-T therapy, etc.) targeting CD19 and CD20, either successively or simultaneously (those who have only received T-cell engaging therapy targeting one of the targets CD19 or CD20can be included).

           25. Use Fredericia's QT correction formula to correct heart rate for QT interval (QTCF)>480msec.

           26. During the dose increase phase, the body weight is less than 40kg. 27. Subjects judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) (Phase I) | Up to 4 weeks
  Number of subjects with a DLT
Maximum tolerated dose (MTD) (Phase I) | Up to 4 weeks
  Determine maximum tolerated dose (MTD) of BR110
Recommended phase 2 dose (RP2D) (Phase I) | Up to 48 weeks
  Determine recommended phase 2 dose (RP2D) of BR110.
Objective response rate (ORR) (Phase II) | Up to 48 weeks
  he primary efficacy outcome is ORR(CR+PR), measured per Lugano 2014 Classification for Lymphomas

SECONDARY OUTCOMES:
Number of subjects with adverse events (Phase Ia) | Up to 48 weeks
  Number of subjects who experienced an adverse event
Pharmacokinetic concentration | Up to 48 weeks
  Describe blood drug concentrations using appropriate statistics based on dose groups and planned time points
Immunogenicity | Up to 48 weeks
  Summarize the number of positive cases and positive rate of ADA by dose group and immunogenicity evaluation time points before and after administration and cumulative positive rate
Disease Control Rate (DCR） | Up to 48 weeks
  Calculate the DCR of each group of subjects at each evaluation time point separately
Progression-Free Survival (PFS) | Up to 48 weeks
  The Kaplan Meier method will be used to calculate the lower quartile (Q1), middle Digits and upper quartile (Q3) and their 95% confidence intervals
Overall Survival (OS) | Up to 48 weeks
  The Kaplan Meier method will be used to calculate the lower quartile (Q1), middle Digits and upper quartile (Q3) and their 95% confidence intervals
The proportion of subjects with CR, PR, SD, PD | Up to 48 weeks
  Calculate the proportion

OTHER OUTCOMES:
Exploratory Objectives(Phase I) | Up to 48 weeks
  Exploring the impact of the production of anti drug antibodies on efficacy and safety
Exploratory Objectives(Phase I) | Up to 48 weeks
  Relationship between dose level causing 100% B-cell depletion in peripheral blood (and PK parameters associated with this) and clinical parameters, including safety and efficacy.
Exploratory Objectives(Phase I) | Up to 48 weeks
  Preliminary exploration of the relationship between pharmacodynamic indicators and efficacy.
Exploratory Objectives(Phase II) | Up to 48 weeks
  To evaluate MRD in NHL patients who achieve a CR using circulating tumor DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China